CLINICAL TRIAL: NCT00843362
Title: A Randomised Controlled Trial of 24-Hours Vaginal Dinoprostone Pessary vs. Gel for Induction of Labour in Term Pregnancies With a Bishop Score ≤4
Brief Title: 24-Hour Vaginal Dinoprostone Pessary Versus Gel for Labour Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Tiziana Frusca, University of Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Spedali Civili 924
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Labor, Induced; Cervical Ripening
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 24-hours vaginal dinoprostone pessary
  Interventions: Drug: Dinoprostone vaginal pessary
- 2 (Active Comparator): Vaginal dinoprostone gel
  Interventions: Drug: Dinoprostone vaginal gel

INTERVENTIONS:
Drug: Dinoprostone vaginal pessary — 10 mg controlled-release dinoprostone pessary applied for 24 hours
  Other Names: Propess, Ferring, Milan, Italy
  Arms: 1
Drug: Dinoprostone vaginal gel — 2 mg vaginal dinoprostone gel, two daily doses with a 6 hours interval
  Other Names: Prepidil, Pharmacia, Milan, Italy
  Arms: 2

SUMMARY:
The aim of induction of labour is to initiate labour when maternal and fetal conditions necessitate delivery before the onset of spontaneous contractions. Prostaglandins are widely used for induction of labour, and can be administered orally, vaginally, intracervically, endovenously and by extra-amniotic or intra-amniotic routes. Dinoprostone is one of the synthetic prostaglandins most commonly used to achieve cervical ripening and labour induction, and can be administered as tablets, suppositories, gel (vaginal and intracervical) or as a controlled-release intravaginal pessary. The controlled-release pessary has some potential advantages: a single application is required; the insert is easily administered and can be removed as soon as labour starts or if complications ensue. Studies comparing the dinoprostone vaginal insert to other prostaglandin formulations have shown variable results, probably influenced by drug administration regimens, indications for induction, and cervical conditions of the women. The purpose of this study is to assess the efficacy of the induction of labour using dinoprostone in patients with an unfavourable cervix, and to compare the efficacy and the cost of 24-hours controlled-release dinoprostone pessary and intravaginal dinoprostone gel.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy, fetal cephalic presentation, Bishop score ≤ 4, gestational age 37-42 weeks

Exclusion Criteria:

* premature rupture of the membranes, history of a previous caesarean section,
* maternal clinical contraindications to the administration of prostaglandins,
* fetal malpresentation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2006-12; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
spontaneous vaginal delivery

SECONDARY OUTCOMES:
induction to labour time
induction to delivery time
rate of failed induction
cost per patient
rate of caesarean section for fetal heart rate abnormalities
5 minute Apgar score < 7
arterial cord blood pH <7.1
uterine hyperstimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynaecology, University of Brescia, Brescia, Italy